CLINICAL TRIAL: NCT06035731
Title: Evaluation of the Medical Service by Socio-aesthetics in Oncology
Acronym: RCT-SE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Valence (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RIPH-CHV-13
Record Dates: First submitted 2023-08-29; First posted 2023-09-13 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Cancer of Colon; Cancer, Lung; Cancer, Breast; Cancer Prostate; Cancer Pain; Anxiety Depression
Keywords: SOCIO-AESTHETIC
MeSH Terms: conditions — Colonic Neoplasms; Lung Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Cancer Pain

STUDY DESIGN:
Intervention Model Description: open label, randomized, controlled, multicenter intervention study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A: well-being care performed by SOCIO-AESTHETICS (Experimental): Group A will benefit from 4 sessions of well being care performed by a qualified socio-aesthetics, during 4 consecutive chemotherapy administrations.
  Patients included will have following interventions :
  quality of life: PCQ Pain: EVA Anxiety: HADS
  Interventions: Other: SOCIO-AESTHETICS care
- group B: control (No Intervention): Group B (control) will apply the dermo-cosmetic products themselves (self-care) without intervention of the socio-aesthetician, during 4 consecutive chemotherapy administrations.
  quality of life: PCQ Pain: EVA Anxiety: HADS

INTERVENTIONS:
Other: SOCIO-AESTHETICS care — SOCIO-AESTHETICS well being care performed by qualify person
  Arms: group A: well-being care performed by SOCIO-AESTHETICS

SUMMARY:
the 3-year randomized controlled RCT-SE study aims to investigate Socio-aesthetics well being care on quality of life, pain and anxiety.

The primary objective is to show that socio-aesthetics well being care improves quality of life during cancer treatment, compared to self care administration of dermo-cosmetics products

The secondary objectives are to show that socio-aesthetics well being care significantly reduced anxiety and pain compared to self care administration of dermo-cosmetics products

DETAILED DESCRIPTION:
Socio-aesthetics care is the delivery appropriate beauty care in a population weakened by a physical, psychological and/or social attack.

this well-being care is imperfectly assessed with few data from randomized controlled trials.

The RCT-STudy is a randomized, controlled, multicenter, open label, intervention study that will be conducted among 400 patients treated with chemotherapy for breast, prostate, colon and lung cancer.

Patients will be randomly assigned to one of the two arms of the study according to a 1:1 ratio:

* Group A will benefit from 4 sessions of well being care performed by a qualified socio-aesthetic person, with dermo-cosmetics product defined, during 4 consecutive chemotherapy administrations .
* Group B (control) will apply the same dermo-cosmetics products themselves (self-care) without intervention of socio-aesthetic, during 4 consecutive chemotherapy administrations

  12 Evaluations will be conducted between chemotherapy cure N° 2 and chemotherapy cure N°5:
* Pain assessed by Eva
* Anxiety assessed by HADS
* impact of socio-aesthetics care care , assessed by Patient Centricity Questionnaire (PCQ) (0 -110)

Data will be recorded using an e-CRF. patient will be recruited over 3 years and will be followed up for 3 months.

Hypothesis:

Socio-aesthetics session significantly improves quality of life and reduced pain and anxiety compared to self care administration of dermo-cosmetics products

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* treated with chemotherapy for lung , breast, colon or prostate cancer
* Able to understand, read, and write French,
* Affiliated with a social security scheme,
* Having dated and signed an informed consent.

Exclusion Criteria:

* Unable to be followed for medical, social, family, geographic or psychological reasons for the duration of the study,
* Deprived of their liberty by court or administrative decision,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Patient Centricity Questionnaire (PCQ): Patient reported outcome: impact of supportive care | up to 12 weeks
  Patient Centricity Questionnaire (PCQ): (0-110) higher scores mean better outcome

SECONDARY OUTCOMES:
pain EVA | up to 12 weeks
  EVA (0-10) higher scores mean worse outcome.
Anxiety | up to 12 weeks
  HADS: Hospital Anxiety and Depression Scale (0-42) higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Guillaume, Principal Investigator — CH VALENCE
Locations (3):
- France (3):
  - Centre Antoine Lacassagne, Nice
  - AP HP, Paris
  - Chru Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided